CLINICAL TRIAL: NCT00667576
Title: Late Phase 2 Study of Paricalcitol Injection: Dose-response Study of Paricalcitol Injection in Chronic Kidney Disease Subjects Receiving Hemodialysis With Secondary Hyperparathyroidism (Examination of Initial Dose and Incremental Dose)
Brief Title: Dose-response Study of Paricalcitol Injection in Chronic Kidney Disease Patients Receiving Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Abbott Japan Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M10-309
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2010-04-02 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Kidney Disease on Hemodialysis; Secondary Hyperparathyroidism
Keywords: chronic kidney disease; secondary hyperparathyroidism; hemodialysis; paricalcitol; maxacalcitol
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic | interventions — maxacalcitol; paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Paricalcitol 2 µg ± 1 µg (Experimental): Paricalcitol initial dosage 2 micrograms (µg) with incremental adjustment of 1 µg
  Interventions: Drug: Paricalcitol
- Paricalcitol 2 µg ± 2 µg (Experimental): Paricalcitol initial dosage 2 µg with incremental adjustment of 2 µg
  Interventions: Drug: Paricalcitol
- Paricalcitol 4 µg ± 1 µg (Experimental): Paricalcitol initial dosage 4 µg with incremental adjustment of 1 µg
  Interventions: Drug: Paricalcitol
- Paricalcitol 4 µg ± 2 µg (Experimental): Paricalcitol initial dosage 4 µg with incremental adjustment of 2 µg
  Interventions: Drug: Paricalcitol
- Maxacalcitol 5 or 10 µg ± 2.5 µg (Other): Maxacalcitol initial dosage 5 or 10 µg with incremental adjustment of 2.5 µg
  Interventions: Drug: Maxacalcitol

INTERVENTIONS:
Drug: Maxacalcitol — Study drug was administered 3 times per week (no more frequently than every other day) intravenously immediately before the completion of hemodialysis. The initial dosage was administered for 2 weeks, with subsequent dosage adjustment based on the subject's iPTH, calcium (adjusted), and phosphorus levels every 2 weeks. Total duration of treatment was 12 weeks.
  Arms: Maxacalcitol 5 or 10 µg ± 2.5 µg
Drug: Paricalcitol — Study drug was administered 3 times per week (no more frequently than every other day) intravenously immediately before the completion of hemodialysis. The initial dosage was administered for 2 weeks, with subsequent dosage adjustment based on the subject's iPTH, calcium (adjusted), and phosphorus levels every 2 weeks. Total duration of treatment was 12 weeks.
  Other Names: ABT-358; Zemplar
  Arms: Paricalcitol 2 µg ± 1 µg; Paricalcitol 2 µg ± 2 µg; Paricalcitol 4 µg ± 1 µg; Paricalcitol 4 µg ± 2 µg

SUMMARY:
The purpose of this study was to investigate the initial dose and dose adjustment range for paricalcitol injection in patients with chronic kidney disease on hemodialysis who have secondary hyperparathyroidism.

DETAILED DESCRIPTION:
This multicenter, randomized, open-label trial consisted of 4 dose-adjustment regimens for paricalcitol injection (initial doses and dose adjustment ranges were 2 ± 1 µg, 2 ± 2 µg, 4 ± 1 µg, and 4 ± 2 µg) and 1 maxacalcitol regimen (initial dose and dose adjustment range was 5 µg ± 2.5 µg or 10 µg ± 2.5 µg) as a reference group. Subjects who met the inclusion criteria were randomized equally to 1 of the treatment groups with iPTH values at screening (< 500 pg/mL or ≥ 500 pg/mL) as a dynamic allocation factor. Study drugs were administered 3 times weekly (every other day) from the venous end of the hemodialysis circuit just before completion of the dialysis session. The initial doses were continued for 2 weeks, followed by dose adjustments (increase, maintenance, decrease, suspension, or resumption) by 1 µg or 2 µg units for the paricalcitol groups and by 2.5 µg units for the maxacalcitol group based on iPTH, calcium (adjusted), and phosphorus values every 2 weeks.

Subjects in the paricalcitol groups were to be suspended from treatment if their iPTH value decreased to < 60 pg/mL in accordance with the guidelines proposed by the Japanese Society of Dialysis Therapy for the treatment of secondary hyperparathyroidism in chronic dialysis patients (control goal value of 60-180 pg/mL for iPTH). The dose adjustment criteria based on iPTH values for the maxacalcitol group were set according to the prescribing information for maxacalcitol (suspended when iPTH decreased to ≤ 150 pg/mL).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic kidney disease receiving hemodialysis 3 times a week for at least 3 months prior to obtaining the informed consent and scheduled to be receiving the same hemodialysis during the study period.
* Using dialysate with constant concentration of calcium for 4 weeks prior to obtaining informed consent and phosphate binder with constant dose regimen for 2 weeks prior to obtaining informed consent.
* Intact parathyroid hormone level (iPTH) ≥ 300 pg/mL
* Calcium (adjusted) 8.4-10.2 milligrams/deciliter (mg/dL)
* Phosphorus ≤ 6.5 mg/dL
* Age ≥ 20 years

Exclusion Criteria:

* History of allergic reaction or significant sensitivity to vitamin D or vitamin D related compounds
* Parathyroidectomy or ethanol infusion within past year
* Progressive malignancy or clinically significant hepatic diseases, severe cerebral/cardiovascular diseases, severe hypertension, or uncontrolled diabetes mellitus
* Drug or alcohol abuse within past 6 months
* Taking calcitonin, maintenance intravenous or oral glucocorticoids, cinacalcet, bisphosphonates, selective estrogen-receptor modulator (SERM), vitamin D compounds (other than study drug), or other drugs that may affect calcium or bone metabolism (other than estrogen or progestin, vitamin K2)
* Will need to take chronic dose (≥ 2 consecutive weeks) of cytochrome P450 (CYP3A) inhibitors (e.g., clarithromycin, grapefruit products) or inducers (e.g., carbamazepine, rifampicin)
* Taking aluminum containing products (2 weeks prior to consent)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryotaro Matsuzawa, Study Director — Abbott
Locations (12):
- Japan (12):
  - Tokyo, Metropolis
  - Aichi, Prefecture
  - Chiba, Prefecture
  - Fukuoka, Prefecture
  - Hokkaido, Prefecture
  - Ibaraki, Prefecture
  - Kanagawa, Prefecture
  - Kumamoto, Prefecture
  - Nagano, Prefecture
  - Nagasaki, Prefecture
  - Osaka, Prefecture
  - Saitama, Prefecture

RESULTS

PARTICIPANT FLOW:
Groups:
- Paricalcitol 2 µg ± 1 µg: Paricalcitol initial dosage 2 µg with incremental adjustment of 1 µg
Period: Overall Study
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg | Maxacalcitol 5 or 10 µg ± 2.5 µg
Started | 30 | 31 | 31 | 31 | 30
Completed | 28 | 30 | 29 | 27 | 29
Not Completed | 2 | 1 | 2 | 4 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 1
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Not completed — Missed Visit | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg | Maxacalcitol 5 or 10 µg ± 2.5 µg | Total
Number analyzed (Participants) | 30 | 31 | 31 | 31 | 30 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 19 | 19 | 12 | 87
  >=65 years | 11 | 13 | 12 | 12 | 18 | 66
Age Continuous [Mean (Standard Deviation); unit: years] | 62.1 (11.94) | 60.7 (11.80) | 58.1 (12.35) | 61.5 (11.17) | 64.1 (11.98) | 61.3 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 11 | 14 | 7 | 64
  Male | 12 | 17 | 20 | 17 | 23 | 89
Region of Enrollment [Number; unit: participants]
  Japan | 30 | 31 | 31 | 31 | 30 | 153

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With ≥ 50% Decrease From Baseline in Intact Parathyroid Hormone (iPTH) Serum Level
Time Frame: Baseline to Week 13 (Final Visit)
Population: The efficacy analysis was performed on the full analysis set (FAS). The FAS included all treated patients, except for 1 subject from the paricalcitol 4 ± 2 µg group who discontinued the study without measurement of iPTH after the first drug injection. Missing data were not imputed.
Measure: Number; unit: Percentage of participants
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg | Maxacalcitol 5 or 10 µg ± 2.5 µg
Number analyzed (Participants) | 30 | 31 | 31 | 30 | 30
Percentage of participants | 53.3 | 41.9 | 38.7 | 56.7 | 43.3

2. Other Pre Specified Outcome: Percentage of Subjects With Hypercalcemia
Description: Hypercalcemia was defined as at least 1 adjusted calcium value > 11.5 mg/dL or at least 2 consecutive adjusted calcium values ≥ 11.0 mg/dL
Time Frame: Through Week 13
Population: Safety analysis was performed on the Safety Set, which included all subjects who received at least 1 dose of study drug. Missing data were not imputed.
Measure: Number; unit: Percentage of participants
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg | Maxacalcitol 5 or 10 µg ± 2.5 µg
Number analyzed (Participants) | 30 | 31 | 31 | 31 | 30
Percentage of participants | 30.0 | 48.4 | 45.2 | 58.1 | 30.0

3. Other Pre Specified Outcome: Percentage of Subjects With Hyperphosphatemia
Description: Hyperphosphatemia was defined as at least 2 consecutive phosphorus values ≥ 7.0 mg/dL
Time Frame: Through Week 13
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg | Maxacalcitol 5 or 10 µg ± 2.5 µg
Number analyzed (Participants) | 30 | 31 | 31 | 31 | 30
Percentage of participants | 10.0 | 9.7 | 9.7 | 19.4 | 13.3

4. Secondary Outcome: Mean Change From Baseline in Intact Parathyroid Hormone (iPTH) Level
Time Frame: Baseline to Week 13 (Final Visit)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg | Maxacalcitol 5 or 10 µg ± 2.5 µg
Number analyzed (Participants) | 30 | 31 | 31 | 30 | 30
pg/mL | -233.2 [-313.37 to -153.03] | -260.8 [-366.64 to -154.90] | -178.2 [-246.22 to -110.10] | -211.7 [-309.14 to -114.33] | -236.6 [-311.46 to -161.68]

5. Secondary Outcome: Percentage of Subjects With Intact Parathyroid Hormone (iPTH) ≤ 180 Picograms/Milliliter (pg/mL)
Time Frame: Baseline to Week 13 (Final Visit)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg | Maxacalcitol 5 or 10 µg ± 2.5 µg
Number analyzed (Participants) | 30 | 31 | 31 | 30 | 30
Percentage of participants | 36.7 | 32.3 | 32.3 | 36.7 | 33.3

6. Secondary Outcome: Percentage of Subjects With 2 or More Decreases of ≥ 50% From Baseline in Intact Parathyroid Hormone (iPTH) Level
Time Frame: Through Week 13
Population: The efficacy analysis was performed on the full analysis set (FAS). The FAS included all treated subjects, except for 1 subject from the paricalcitol 4 ± 2 µg group who discontinued the study without measurement of iPTH after the first drug injection. Missing data were not imputed.
Measure: Number; unit: Percentage of participants
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg | Maxacalcitol 5 or 10 µg ± 2.5 µg
Number analyzed (Participants) | 30 | 31 | 31 | 30 | 30
Percentage of participants | 90.0 | 100 | 90.3 | 90.0 | 93.3

7. Secondary Outcome: Duration of 2 Consecutive Decreases of ≥ 50% From Baseline in Intact Parathyroid Hormone (iPTH) Values
Time Frame: Through Week 13
Population: Includes subjects from the Full Analysis Set (FAS) who had 2 consecutive iPTH decreases of ≥ 50% from baseline. Missing data were not imputed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg | Maxacalcitol 5 or 10 µg ± 2.5 µg
Number analyzed (Participants) | 27 | 30 | 28 | 27 | 28
days | 23.8 (14.34) | 27.7 (14.60) | 29.0 (15.26) | 25.2 (18.21) | 10.9 (12.18)

8. Secondary Outcome: Duration of 2 Consecutive Intact Parathyroid Hormone (iPTH) Values ≤ 180 pg/mL
Time Frame: Through Week 13
Population: Includes subjects from the Full Analysis Set (FAS) who had 2 consecutive iPTH values ≤ 180 pg/mL. Missing data were not imputed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg | Maxacalcitol 5 or 10 µg ± 2.5 µg
Number analyzed (Participants) | 20 | 25 | 24 | 22 | 23
days | 22.0 (12.23) | 26.1 (15.36) | 19.7 (13.32) | 17.2 (15.52) | 3.1 (3.29)

ADVERSE EVENTS:
Time Frame: Adverse events were collected after the first dose of study drug until 30 days after the last dose of study drug (up to 12 weeks of treatment).
Description: The investigator recorded any undesirable medical events (adverse events) during the study period based on medical interview of the subject, information from medical staff, or spontaneous reporting by the subject.
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg | Maxacalcitol 5 or 10 µg ± 2.5 µg
Serious Adverse Events (participants affected / at risk) | 1/30 | 2/31 | 3/31 | 2/31 | 2/30
Other Adverse Events (participants affected / at risk) | 30/30 | 29/31 | 30/31 | 28/31 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol 2 µg ± 1 µg (N=30) | Paricalcitol 2 µg ± 2 µg (N=31) | Paricalcitol 4 µg ± 1 µg (N=31) | Paricalcitol 4 µg ± 2 µg (N=31) | Maxacalcitol 5 or 10 µg ± 2.5 µg (N=30)
shunt stenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
shunt aneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
cerebellar infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
iliac artery stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
arteriosclerosis obliterans (Vascular disorders) | 0 | 0 | 0 | 1 | 0
femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol 2 µg ± 1 µg (N=30) | Paricalcitol 2 µg ± 2 µg (N=31) | Paricalcitol 4 µg ± 1 µg (N=31) | Paricalcitol 4 µg ± 2 µg (N=31) | Maxacalcitol 5 or 10 µg ± 2.5 µg (N=30)
abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 1
cheilitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
constipation (Gastrointestinal disorders) | 2 | 4 | 1 | 1 | 2
dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
diarrhea (Gastrointestinal disorders) | 3 | 3 | 2 | 1 | 0
epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
puncture site haemorrhage (General disorders) | 0 | 2 | 0 | 0 | 0
hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 2
nasopharyngitis (Infections and infestations) | 9 | 9 | 10 | 9 | 9
pharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 1
upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 1 | 0
arthropod sting (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 2
contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 4
fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 3
procedural hypotension (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2 | 1
shunt occlusion (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 0 | 1
wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
blood pressure decreased (Investigations) | 0 | 0 | 0 | 2 | 0
hypercalcaemia (Metabolism and nutrition disorders) | 12 | 19 | 20 | 23 | 13
hyperphosphataemia (Metabolism and nutrition disorders) | 6 | 10 | 6 | 12 | 8
arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 0 | 1
back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 3
muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 1
myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 3
headache (Nervous system disorders) | 0 | 3 | 2 | 3 | 0
restless leg syndrome (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 1
pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 2 | 4
skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0
hypertension (Vascular disorders) | 1 | 6 | 1 | 3 | 4

LIMITATIONS AND CAVEATS:
Different PTH thresholds were applied for suspending study drug: paricalcitol groups <60 pg/mL, maxacalcitol group ≤150 pg/mL. This study was not statistically powered to compare treatments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.